CLINICAL TRIAL: NCT01281878
Title: PILOTSTUDIE ZUR PYRIDOXALPHOSPHATTHERAPIE BEI PATIENTEN MIT PRIMÄRER HYPEROXALURIE TYP I (PHOX-B6-PILOT) Pilot Trial on Treatment of Patients With Primary Hyperoxaluria Type I With Pyridoxal-phosphate
Brief Title: Trial on Treatment of Patients With Primary Hyperoxaluria Type I With Pyridoxal-phosphate
Acronym: PHOX-B6-Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. B. Hoppe, Prof. Dr. med. Bernd Hoppe, University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1251
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Primary Hyperoxaluria Type I
Keywords: primary hyperoxaluria; Pyridoxal-phosphate
MeSH Terms: conditions — Hyperoxaluria; Hyperoxaluria, Primary | interventions — Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyridoxal-phosphate (Experimental): Treatment with pyridoxal-phosphate in increasing dosages every six weeks starting with 5mg/kg body weight up to 20 mg/kg body weight. treatment duration 24 weeks
  Interventions: Drug: Vitamin B 6

INTERVENTIONS:
Drug: Vitamin B 6 — Oral solution of pyridoxal phosphate start with 5mg per kg body weight per day in two dosages over 6 weeks, increase stepwise by 5mg/kg body weight every 6 weeks up to 20 mg/kg body weight/d.

SUMMARY:
In this study the investigators will prospectively analyze the reduction of urinary oxalate excretion under the treatment with PLP in dosages of 5mg/kg/day up to 20 mg/kg/day and serum level response relationship with PLP as an i.v. solution used orally in 12 patients with primary hyperoxaluria type I as an inherited autosomal-recessive-disorder leading to increased endogenous oxalate production, urolithiasis and end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of diagnosis of PH I by any one of the following:

  * Liver biopsy confirmation of deficient liver specific peroxisomal alanine-glyoxylate aminotransferase, (AGT or mislocalization of AGT from peroxisomes to mitochondria)
  * Homozygosity or compound heterozygosity for a known mutation in the causative gene (AGXT) for PH I
* Male or female subjects between 5 years and 60 years of age
* Renal function defined as an estimated GFR > 60 ml/min normalized to 1.73 m2 body surface area
* Subjects receiving pyridoxal-phosphate before the study must be willing to discontinue therapy with pyridoxal-phosphate for a wash out phase of at least 4 weeks but always until normalization of serum pyridoxal-phosphate levels
* Written informed consent from patients and/or legally acceptable representatives

Exclusion Criteria:

* Pregnant or lactating women
* Women of child-bearing potential who are not using a highly effective contraception method with a pearl-index < 1. Highly effective contraception methods are oral, transdermal, injectable, or implanted contraceptives, IUD, abstinence, or sterile sexual partner and must agree to continue using such precautions during the pyridoxal-phosphate study
* Subjects post liver or kidney transplantation or combined transplantation
* Chronic diarrhoea with the risk of malabsorption
* Any other abnormal finding such as physical examination or laboratory evaluation, in the opinion of the investigator, is indicative of a disease that would compromise the safety taking pyridoxal-phosphate per os and the absorption
* Subjects participating in other clinical trials with investigational products 4 weeks prior to trial entry, during the trial and 4 weeks after the trial
* Subjects who are unable to take the trial medication
* Subjects who are unable to collect 24-hour urine samples or follow other study procedures
* Subjects who are under treatment with L-Dopa, Isoniazid, D-Penicillamine (interactions between these drugs and pyridoxal-phosphate are known and might influence serum pyridoxal-phosphate levels)
* Subjects with known allergies to substances of contents (e.g. Potassium sorbet, raspberry syrup)
* Subjects confined to an institution on judicial or official behalf
* Subjects who are in dependency to the sponsor or the PI of the trial

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the reduction of the urinary oxalate excretion (percentage change in urinary oxalate, expressed as mmol/1.73 m2 /day) at week 24 compared to baseline. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Children´s Hospital University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Hoyer-Kuhn H, Kohbrok S, Volland R, Franklin J, Hero B, Beck BB, Hoppe B. Vitamin B6 in primary hyperoxaluria I: first prospective trial after 40 years of practice. Clin J Am Soc Nephrol. 2014 Mar;9(3):468-77. doi: 10.2215/CJN.06820613. Epub 2014 Jan 2. PMID 24385516